CLINICAL TRIAL: NCT00527878
Title: A Double-Blind, Randomized, Placebo-Controlled Cross-Over Study Assessing the Role of Pathogen-Specific IgE and Histamine Release in the Hyper-IgE Syndrome and the Effect of Ranitidine on Laboratory and Clinical Manifestations
Brief Title: Effect of Ranitidine on Hyper-IgE Recurrent Infection (Job's) Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to enroll adequate patient numbers due to small number of eligible patients
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Steven M. Holland, M.D./National Institute of Allergy and Infectious Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 070218; 07-I-0218
Record Dates: First submitted 2007-09-08; First posted 2007-09-11 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: JOB's Syndrome; Hyper-IgE Recurrent Infection Syndrome; Immune Deficiency
Keywords: Hyper-IgE Recurrent Infection Syndrome; Ranitidine Therapy; Job's Syndrome; Cross-Over Study; Double-Blind Placebo Controlled; Hyper-IgE Syndrome; Job Syndrome; Immune Deficiency
MeSH Terms: conditions — Job Syndrome; Immunologic Deficiency Syndromes | interventions — Ranitidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo/Ranitidine crossover (Experimental): Patients took placebo for 12 months and then ranitidine for 12 months
  Interventions: Drug: Ranitidine; Drug: Placebo
- Ranitidine/placebo crossover (Experimental): Ranitidine for one year followed by placebo for one year
  Interventions: Drug: Ranitidine; Drug: Placebo

INTERVENTIONS:
Drug: Ranitidine — Double blinded, randomized placebo controlled crossover study. Patients received 12 months of placebo and 12 months of treatment medication (ranitidine).
Drug: Placebo

SUMMARY:
This study will examine the safety and effectiveness of ranitidine (Zantac) in patients with Hyper-IgE recurrent infection syndrome, a disease characterized by recurrent infections of the ears, sinuses, lungs and skin, and abnormal levels of the antibody immunoglobulin E (IgE).

Patients age 2 and older who have Hyper-IgE recurrent infection syndrome and who have had chronic or frequent infections in the last 12 months may be eligible for this study.

Participants are randomly assigned to take ranitidine or placebo in pill or liquid form twice a day for 12 months. In addition to treatment, patients undergo the following procedures during visits scheduled on day 0 of the study (baseline) and at 3, 12, 15 and 24 months. Evaluations at 6, 9, 18 and 21 months are by telephone.

* Medical history and physical examination - baseline and 3 and 24 months.
* Clinical severity score - baseline and 3, 6, 9, 12, 15, 18, 21 and 24 months.
* Dermatology exam - baseline and 3, 12, 15 and 24 months.
* Pulmonary function test - baseline and 12 and 24 months.
* Chest CT - baseline and 12 and 24 months.
* Quality of life assessment - baseline and 3, 12, 15 and 24 months.
* Pregnancy testing - baseline and 3, 12, 15 and 24 months.
* HIV test - baseline and 12 and 24 months.
* Contraception evaluation - baseline and 3, 6, 9, 12, 15, 18, 21 and 24 months.
* Missed school/work days assessment - baseline and 3, 12, 15 and 24 months.
* Medication adherence - baseline and 3, 6, 9, 12, 15, 18, 21 and 24 months.

In addition to the above procedures, participants who are not enrolled in study 00-I-0159 have a baseline scoliosis series and genetic consult.

DETAILED DESCRIPTION:
Hyper-immunoglobulin E (IgE) syndrome (HIES) is a rare primary immunodeficiency characterized by eczema, recurrent skin and lung infections, elevated serum IgE, and multiple connective tissue and skeletal abnormalities. The autosomal dominant form of HIES is caused primarily by a mutation in the STAT3 gene. Patients with HIES produce IgE antibodies specific for Candida albicans and Staphylococcus aureus, two of the common pathogens in this population. We hypothesize that the presence of pathogen-specific IgE, combined with continuous exposure to these ubiquitous agents, leads to chronic IgE-mediated histamine release from basophils and mast cells, with subsequent pathogen-specific immune tolerance and an increase in pathogen-specific T regulatory cells. We plan to test this hypothesis through clinical and immunologic evaluation of HIES patients before, during, and after histamine-2 receptor (H2) blocker therapy with ranitidine through a prospective, placebo-controlled crossover study. We chose this therapy because histamine has been shown to stimulate interleukin-10 (IL-10), a major down regulatory cytokine, through the H2 receptor, and clinical improvement has been observed in several patients treated with H2 blockers. Laboratory studies will include determinations of pathogen-specific immunoglobulin G4 (IgG4):IgE ratios, basophil activation, IL-10 producing regulatory T-cells, cellular proliferative responses to staphylococcal and candidal antigens, and functional testing of regulatory T-cells. Clinical evaluations will include comprehensive history and physical examination, dermatologic evaluation, genetic evaluation for clinical severity scoring of HIES, pulmonary function tests, and chest computerized tomography (CT) examination. Through this study, we will further our understanding of the immunologic abnormalities of HIES and determine whether a larger prospective, double-blind trial of H2 blockade as adjunctive therapy for HIES is indicated.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male and female patients with the diagnosis of Hyper IgE Recurrent Infection (Job) syndrome. Mutations in the STAT3 gene account for the majority, if not all cases of HIES. However as the full genetics of HIES remains unknown, we will use clinical criteria, including the expert opinion of the investigators, as well as a score greater than 40 by the diagnostic scoring system used in protocol 00-I-0159.
  2. A chronic (greater than 4 weeks duration) infection or greater than 2 acute infections within the last 12 months. Acute infections can include but are not limited to: pneumonia, abscesses, sinusitis, skin infections, mucocutaneous candidiasis and ear infections. Chronic infections include continuous or intermittent symptoms despite appropriate therapeutic interventions for at least 4 weeks, including but not limited to chronic lung infiltrates with productive cough, chronic ear drainage despite topical therapy, chronic or intermittent drainage from a single abscess site, and/or chronic signs of sinusitis on sinus CT scan.
  3. Patients aged 2 years and above. There is no upper age limit. We are excluding children less than 2 years of age, as we do not expect them to meet the first inclusion criterion, having a score high enough to be diagnosed with HIES.
  4. Patients have to be at their own personal clinical baseline for at least 2 weeks duration. Patients will not start the study medication during an acute exacerbation of and infection.
  5. The patient or the patient's guardian will be willing and capable of providing informed consent after initial counseling by clinical staff. Separate consent forms for all interventional procedures will be obtained after explanation of the specific procedure.
  6. Patients must agree to have blood stored for future studies of the immune system and/or other medical conditions.
  7. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
  8. Patients may be concurrently enrolled on other protocols as long as the Principal Investigator (PI) is informed.

EXCLUSION CRITERIA:

1. Pregnancy. Ranitidine is pregnancy class B, and likely safe in pregnancy, but as this has not been studied, pregnant patients will be excluded. In addition, hormonal changes that occur during pregnancy may affect the skin manifestations and frequency of infection.
2. Hypersensitivity to ranitidine or any of the ingredients in ranitidine.
3. Pre-existing medications or conditions for which the investigators judge that ranitidine should not be given.
4. Patient or investigators unwilling to stop baseline H2 receptor antagonist therapy (over the counter or prescription) such as Tagamet (Cimetidine), Pepcid (Famotidine), and Axid (Nizatidine). H2 receptor antagonist therapy must be stopped for 3 months prior to study initiation. Patients who are receiving H2 receptor antagonist therapy for gastritis, acid reflux, or peptic ulcer disease will be offered changing their regimen to a proton pump inhibitor or other non-H2 receptor antagonist therapy to allow for study enrollment (3 months after stopping the H2 receptor antagonist).
5. Patients under the age of 2 years
6. Patients with HIV, receiving chemotherapy or who have a malignancy.
7. Any condition that in the judgment of the investigator would place the subject at undue risk or compromise the results or interpretation of the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Grimbacher B, Holland SM, Gallin JI, Greenberg F, Hill SC, Malech HL, Miller JA, O'Connell AC, Puck JM. Hyper-IgE syndrome with recurrent infections--an autosomal dominant multisystem disorder. N Engl J Med. 1999 Mar 4;340(9):692-702. doi: 10.1056/NEJM199903043400904. PMID 10053178
- [Background] Davis SD, Schaller J, Wedgwood RJ. Job's Syndrome. Recurrent, "cold", staphylococcal abscesses. Lancet. 1966 May 7;1(7445):1013-5. doi: 10.1016/s0140-6736(66)90119-x. No abstract available. PMID 4161105
- [Background] Buckley RH, Wray BB, Belmaker EZ. Extreme hyperimmunoglobulinemia E and undue susceptibility to infection. Pediatrics. 1972 Jan;49(1):59-70. No abstract available. PMID 5059313

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 participants were screened but only 14 participants were randomized. Two individuals decided not to participate.
Groups:
- Placebo/Ranitidine: Ranitidine will be dosed orally at 150 mg twice daily for adults, and at 2-4 mg/kg/dose twice daily for children with a maximum dose of 150 mg twice daily. Liquid formulations will be provided for individuals unable to swallow pills. Subjects will be randomized to receive placebo for 12 months followed by 12 months of the ranitidine.
- Ranitidine/Placebo: Ranitidine will be dosed orally at 150 mg twice daily for adults, and at 2-4 mg/kg/dose twice daily for children with a maximum dose of 150 mg twice daily. Liquid formulations will be provided for individuals unable to swallow pills. Subjects will be randomized to receive ranitidine for 12 months followed by 12 months of the ranitidine.
Period: Intervention 1
Arm/Group | Placebo/Ranitidine | Ranitidine/Placebo
Started | 7 | 7
Completed | 5 | 4
Not Completed | 2 | 3
Period: Intervention 2
Arm/Group | Placebo/Ranitidine | Ranitidine/Placebo
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants whether or not they were randomized.
Arm/Group | Patients
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 10
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Infections in Subjects With HIES.
Description: Patients received one year of treatment medication and one year of placebo. New infections (bacterial, fungal, viral or parasitic) were defined as those requiring an addition or change of an antimicrobial (including topical, oral or intravenous therapies) or those requiring a medical procedure (i.e., incision and drainage of a skin abscess, warm soaks to aid abscess drainage or sinus drainage).
Time Frame: 1 year on intervention
Population: Patients that completed both arms of the study (24 months)
Measure: Median (Full Range); unit: infections
Groups:
- Placebo: Crossover study in which patients received one year of placebo and one year of ranitidine. This analysis will include the placebo for both arms.
- Ranitidine: Crossover study in which patients received one year of placebo and one year of ranitidine. This analysis will include the treatment for both arms.
Arm/Group | Placebo | Ranitidine
Number analyzed (Participants) | 9 | 9
infections | 4 [2 to 25] | 4 [0 to 15]

2. Secondary Outcome: New Skin Infections
Description: Patients reported the number of new skin infections
Time Frame: 12 months placebo/12 months ranitidine
Population: Patients that completed the study
Measure: Median (Full Range); unit: skin infections
Arm/Group | Placebo | Ranitidine
Number analyzed (Participants) | 9 | 9
skin infections | 1 [0 to 14] | 0 [0 to 10]

3. Secondary Outcome: New Lung Infections
Description: Number of new infection while on placebo or study drug
Time Frame: 12 months placebo and 12 months ranitidine
Population: Patients who completed the study
Measure: Median (Full Range); unit: new lung infections
Arm/Group | Placebo | Ranitidine
Number analyzed (Participants) | 9 | 9
new lung infections | 1 [0 to 4] | 0 [0 to 4]

4. Secondary Outcome: Clinical Severity Score
Description: Scoring that was completed every 3 months. Clinical severity scored had outcomes that could range from 0 to 121 with 0 being the least severe and 121 being the most severe.
Time Frame: one year on ranitidine and one year on placebo
Population: Patients who completed the study
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Ranitidine
Number analyzed (Participants) | 9 | 9
score on a scale | 9.8 [3.2 to 27.5] | 8.5 [3.5 to 30.3]

ADVERSE EVENTS:
Description: Adverse events were not analyzed for each participant as 7 participants did not complete the study and so we were not able to evaluate for adverse events for both placebo and study medication.
Groups:
- Placebo: this was a crossover study and patients received both placebo and study drug (ranitidine), both of which for 12 months, unless they terminated the study.
- Ranitidine: This was a crossover study and patients received 12 months of ranitidine and 12 months of placebo, unless they terminated the study.
Arm/Group | Placebo | Ranitidine
Serious Adverse Events (participants affected / at risk) | 4/11 | 4/12
Other Adverse Events (participants affected / at risk) | 10/11 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | Ranitidine (N=12)
asthma (Respiratory, thoracic and mediastinal disorders) | 0 (1) | 1 — Not thought to be related
hypotension (Cardiac disorders) | 1 | 0 — Not thought to be related to study
pneumonia (Infections and infestations) | 1 | 0 — Thought to be related to underlying disease
pneumonia (Infections and infestations) | 0 | 1 — Thought to be related to underlying study
skin abscess (Infections and infestations) | 1 | 0 — thought to be related to underlying disease
groin abscess (Infections and infestations) | 0 | 1 — thought to be related to underlying disease
central line infection (Infections and infestations) | 1 | 0 — Not thought to be related to study medication
death from respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — patient with death presumed to be related to narcotics.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | Ranitidine (N=12)
sinusitis (Infections and infestations) | 4 | 6
otitis (Infections and infestations) | 4 | 4
upper respiratory tract infection (Infections and infestations) | 4 | 5
gastric ulcer (Gastrointestinal disorders) | 1 | 0
anemia (Blood and lymphatic system disorders) | 3 | 1
neutropenia (Blood and lymphatic system disorders) | 3 | 4
cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
abscess (Infections and infestations) | 4 | 5
chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
pruritus (Immune system disorders) | 1 | 2
vomiting (Gastrointestinal disorders) | 1 | 2
Streptococcal sore throat (Infections and infestations) | 0 | 1
rash (Skin and subcutaneous tissue disorders) | 2 | 3
arthralgias (Musculoskeletal and connective tissue disorders) | 0 | 1
elevated alkaline phosphatase (Hepatobiliary disorders) | 2 | 0
candidiasis (Infections and infestations) | 2 | 2
fever (Infections and infestations) | 2 | 1
folliculitis (Skin and subcutaneous tissue disorders) | 0 | 1
nausea (Gastrointestinal disorders) | 2 | 1
Dental problems (General disorders) | 1 | 1
abdominal pain (Gastrointestinal disorders) | 1 | 1
pain (General disorders) | 0 | 1
tongue ulcer (General disorders) | 1 | 0
pneumonia (Infections and infestations) | 2 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
elevated Liver function tests (Hepatobiliary disorders) | 1 | 1
occult blood in stool (Gastrointestinal disorders) | 1 | 0
eyelid stye (Eye disorders) | 1 | 1
infection (Infections and infestations) | 1 | 0
urinary tract infection (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No